CLINICAL TRIAL: NCT06562803
Title: Efficacy and Safety of Double Plasma Cytokine Adsorption System With Sequential Low-Dose Plasma Exchange in Treating Acute-on-Chronic Liver Failure and Sepsis: A Randomized Controlled Study
Brief Title: Efficacy and Safety of Cytokine Adsorption and Plasma Exchange in Patients With ACLF and Sepsis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Liang Peng, Professor, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PL18
Record Dates: First submitted 2024-08-15; First posted 2024-08-20 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Acute-On-Chronic Liver Failure; Sepsis
MeSH Terms: conditions — Acute-On-Chronic Liver Failure; Sepsis | interventions — Plasma Exchange

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Double plasma cytokine adsorption system with sequential low-dose plasma exchange (Experimental): 30 patients in this group will receive treatment of double plasma cytokine adsorption system with sequential low-dose plasma exchange (DPCAS+LPE) and comprehensive internal medical treatment.
  Interventions: Device: double plasma cytokine adsorption system with sequential low-dose plasma exchange
- Plasma exchange (Active Comparator): 30 patients in this group will receive treatment of plasma exchange(PE) and comprehensive internal medical treatment.
  Interventions: Other: plasma exchange

INTERVENTIONS:
Device: double plasma cytokine adsorption system with sequential low-dose plasma exchange — Both groups received comprehensive medical treatment, including antiviral therapy, anti-infection treatment, supportive care, symptomatic treatment, and prevention of complications. Artificial liver therapy was initiated for both groups on the day of enrollment, with treatments administered every other day for a total of three sessions.
  The experimental group： The first two sessions consisted of a double plasma cytokine adsorption system with sequential low-dose plasma exchange (DPCAS+LPE). This involved using a cytokine adsorption column (CA280,Jafron Biomedical Co., Ltd., Zhuhai, China) and a bilirubin adsorption device (BS330,Jafron Biomedical Co., Ltd., Zhuhai, China) on the same treatment circuit. DPCAS treatment was performed first, with an adsorption volume of 4500ml to 5000ml over 2 to 3 hours, followed by plasma exchange (PE), with 1000ml of plasma and 500ml of 4% albumin being infused. The third treatment was plasma exchange, with the same dosing as in the control group.
  Arms: Double plasma cytokine adsorption system with sequential low-dose plasma exchange
Other: plasma exchange — Based on comprehensive medical treatment, the control group received plasma exchange(PE) treatment, where whole blood was processed through a plasma separator (MICROPLAS MPS 07, BELLCO S.R.L., Italy), with a portion of the plasma discarded and replaced with 1000ml of plasma and 500ml of 4% albumin.Three sessions of plasma exchange (PE) performed every other day.
  Arms: Plasma exchange

SUMMARY:
This study aims to evaluate the efficacy and safety of the double plasma cytokine adsorption system with sequential low-dose plasma exchange (DPCAS+LPE) in patients with acute-on-chronic liver failure (ACLF) complicated by sepsis. The focus is on assessing the impact of the cytokine adsorption column(CA280,Jafron Biomedical Co., Ltd., Zhuhai, China) on survival rates, inflammation markers, and organ function to determine its potential value in clinical practice.

The primary research questions are: (1) Does DPCAS+LPE artificial liver therapy improve the 4-week mortality rate in ACLF patients with sepsis? (2) Does it improve the 12-week mortality rate in these patients? Additionally, the study examines the effects of this therapy on APACHE II scores, SOFA scores, vasoactive-inotropic score, MELD scores, and COSSH-ACLF II scores, as well as the cytokine adsorption efficiency of the CA280.

Patients were randomly assigned to either the DPCAS+LPE group or the plasma exchange(PE) group. All patients received artificial liver therapy every other day, for a total of two sessions. Follow-up assessments were conducted before and after each therapy session, as well as at 1, 2, 3, 4, and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 65 years.
2. Total bilirubin (TBIL) > 12 mg/dL, 3.5>INR ≥ 1.5.
3. Meets the diagnostic criteria for sepsis 3.0: confirmed or suspected infection with an increase in SOFA score by ≥ 2 points.
4. High inflammatory state: IL-6 > 80 pg/ml.
5. Onset of sepsis within the past 72 hours.

Exclusion Criteria:

1. Presence of genetic metabolic liver disease.
2. Patients with liver malignancies or other concurrent cancers.
3. Pregnancy or lactation.
4. Patients with HIV infection or other immunodeficiency diseases.
5. Patients with autoimmune diseases, recent cardiovascular events leading to unstable infarction, or a history of organ transplantation.
6. End-stage organ failure:

   End-stage chronic obstructive pulmonary disease, end-stage pulmonary heart disease, brain death, or persistent vegetative state, Grade IV hepatic encephalopathy.

   End-stage renal disease or acute renal failure requiring CRRT. Inability to maintain a mean arterial pressure above 65 mmHg despite adequate fluid resuscitation, vasopressors, and steroid therapy.
7. Platelet count < 50×10⁹/L, severe coagulopathy, or active bleeding.
8. Allergic reactions to extracorporeal circulation, hemoperfusion substances, or history of severe allergies.
9. Inability to comply with study protocols or refusal to sign the informed consent form.
10. Inability to attend regular follow-up visits according to the study schedule.
11. Any other conditions that, in the investigator's judgment, make the patient unsuitable for inclusion in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-27 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Mortality rate | 4 weeks
  4-week mortality rate

SECONDARY OUTCOMES:
Mortality rate | 12 weeks
  12-week Mortality rate
Changes in Acute Physiology and Chronic Health Evaluation II score from baseline | 1, 2, 3, and 4 weeks
  The theoretical maximum value of Acute Physiology and Chronic Health Evaluation II score（APACHE II score） was 71 points. The higher the score, the higher the risk of death. Patients with more than 15 points were classified as severe, and patients with less than 15 points were classified as non-severe.
Changes in sequential organ failure assessment score from baseline | 1, 2, 3, and 4 weeks
  The theoretical value range of sequential organ failure assessment（SOFA） score is 6-24. The higher the score, the worse the prognosis.
Changes in vasoactive-inotropic score from baseline | 1, 2, 3, and 4 weeks
  Vasoactive-Inotropic Score ( VIS ) evaluates cardiac function and the intensity of vasoactive drug therapy in critically ill patients by quantifying the dose of vasoactive and inotropic drugs received by patients. VIS has no special value range. The higher the score, the higher the patient 's dependence on vasoactive drugs.
Changes in Model for End-Stage Liver Disease score from baseline | 1, 2, 3, and 4 weeks
  MELD score is now widely used in the prioritization of liver transplantation candidates in many countries. The score range is usually between 6 ( low risk ) and 40 ( high risk ).
Changes in COSSH-ACLF II score from baseline | 1, 2, 3, and 4 weeks
  COSSH-ACLF II is a prognostic scoring system for hepatitis B virus -related acute-on-chronic liver failure（HBV-ACLF）. COSSH-ACLF IIs can significantly divide ACLF patients into three risk groups based on two cutoff values of 7.4 and 8.4 : low-risk group ( < 7.4 points ), medium-risk group ( 7.4-8.4 points ) and high-risk group ( ≥ 8.4 points ).
Adsorption rates of various cytokines | Day2, Day4
  Adsorption rates of various cytokines (including pro-inflammatory and anti-inflammatory cytokines) after each treatment
Adsorption rates of lactate | Day2, Day4
  Adsorption rates of lactate after each treatment

CONTACTS AND LOCATIONS:
Overall Officials: Liang Peng, Doctor, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
The study protocol, results and conclusions of this clinical trial will be published at academic conferences or in journals.
Supporting Information: Study Protocol, CSR
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Proposals should be directed to pliang@mail.sysu.edu.cn. To gain access, data requestors will need to sign a data access agreement.